CLINICAL TRIAL: NCT07215260
Title: The Effect of BI 3000202 on the Pharmacokinetics of Rosuvastatin and Digoxin Given as a Cocktail - an Open-label, Non-randomised, 2-period Fixed-sequence Trial in Healthy Male and Female Trial Participants
Brief Title: A Study in Healthy People to Test Whether BI 3000202 Affects How 2 Other Medicines (Rosuvastatin and Digoxin) Are Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1509-0014; 2025-520656-29-00 (Registry Identifier: CTIS); U1111-1317-7517 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-10-09; First posted 2025-10-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Intervention Model Description: Participants cross over from reference treatment (R) to test treatment (T) (two periods, fixed sequence).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cocktail (Reference) then BI 3000202-Cocktail (Test) (Experimental): Cocktail consisting of rosuvastatin and digoxin.
  Interventions: Drug: BI 3000202; Drug: Rosuvastatin; Drug: Digoxin

INTERVENTIONS:
Drug: BI 3000202 — BI 3000202
Drug: Rosuvastatin — Rosuvastatin
  Other Names: CRESTOR®
Drug: Digoxin — Digoxin
  Other Names: Lanicor®

SUMMARY:
The objective of this trial is to assess the effect of BI 3000202 on the pharmacokinetics of rosuvastatin and digoxin given as a cocktail.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure BP, pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg / m^2 (inclusive)
* Signed and dated written informed consent in accordance with international council for harmonisation-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial
* Further inclusion criteria apply.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-11-05 (Actual); Primary Completion 2025-12-07 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 7
Area under the concentration-time curve of digoxin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 7
Maximum measured concentration of rosuvastatin in plasma (Cmax) | Up to Day 7
Maximum measured concentration of digoxin in plasma (Cmax) | Up to Day 7

SECONDARY OUTCOMES:
Area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to Day 7
Area under the concentration-time curve of digoxin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com